CLINICAL TRIAL: NCT04943107
Title: Effect of Antihypertensive Drugs on Glaucoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0287
Record Dates: First submitted 2021-06-16; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy control: adults without glaucoma history or hypertension history
  Interventions: Other: no intervention
- glaucoma patients: adults with primary glaucoma history; without glaucoma-related operation history; without hypertension history
  Interventions: Other: no intervention
- hypertension patients: adults with primary hypertension history; without glaucoma history
  Interventions: Other: no intervention
- glaucoma+hypertension: adults with primary glaucoma history and primary hypertension history; without glaucoma-related operation history
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention, only measurement of blood pressure, intraocular pressure, hypertensive history questionnaire, retinal imaging, optical coherence tomography examination etc..

SUMMARY:
It has been reported that among Asian non-glaucomatous, antihypertensive medications were associated with retinal nerve fiber layer and ganglion cell-inner plexiform layer thickness. In order to explore whether antihypertensive medications would influence the neuropathy among glaucomatous population, we designed a cross-sectional observational study to analyze the retinal status among glaucoma patients with use of antihypertensive medication.

DETAILED DESCRIPTION:
we designed a cross-sectional obeservational study to analyze the retinal status among glaucoma patients with use of hyertensive medication.

ELIGIBILITY:
Inclusion Criteria:

* age no less than 18 years

  * best corrected visual acuity better than decimal 0.3

Exclusion Criteria:

* secondary glaucoma

  * secondary hypertension
  * glaucoma-related operation history
  * pregnancy or lactation period
  * uncooperative with retinal examination
  * severe opacity with refracting media in eye
  * severe retinal diseases and neuropathy
  * congenital retinal optic nerve abnormality
  * other systemic diseases that influence hypertension and glaucoma assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient from ophthalmology and cardiology clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
retinal nerve fiber layer thickness | within 3 months from recruitment
  retinal nerve fiber layer thickness measured by optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Kaijun Wang, MD, Principal Investigator — Second Affiliated Hospital of College of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China